CLINICAL TRIAL: NCT01428609
Title: Blood Mercury Levels Following Retrograde Amalgam Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Masoud Saatchi (Other)
Collaborators: Isfahan University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Masoud Saatchi, Associate Professor of Endodontics, Isfahan University of Medical Sciences
Organization: Isfahan University of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Triple
Other Study IDs: MUI79275
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Blood Mercury Concentration
Keywords: Amalgam; Mercury; Endodontics; Apicoectomy
MeSH Terms: interventions — Dental Amalgam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Amalgam — In all surgical intervention a zinc free amalgam (Tytin. Kerr Sybron Crop., Romulus, MI) was used in the root end prepared spaces as root end filling material. Blood samples were collected in three period of time immediately before and immediately after each surgery and also one week later.
  Other Names: cold-vapor atomic absorption spectrometry(Shimadzu, AA-10)

SUMMARY:
The aim of this study is to determine the blood's mercury level of patients who had amalgam root end filling surgeries. It is to be examined if the mercury concentration in blood is elevated by using amalgam retroseal.

DETAILED DESCRIPTION:
* A total of 14 patients who needs surgical root canal therapy (SRCT) participated in this clinical study.
* The Isfahan University Human Subjects Review Committee approved the protocol of the study.
* All patients filled in the consent form.
* Apicoectomy with retrograde amalgam filling performed for all participant.
* Blood samples were collected in three period of time immediately before and immediately after each surgery and also one week later.
* Each time 10 ml blood was drawn from each patient.
* Analysis of total mercury in blood samples was performed using cold-vapor atomic absorption spectrometry

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* without physician-diagnosed psychological, behavioral, neurological, immunosuppressive, or renal disorders
* having a tooth that required apical surgery

Exclusion Criteria:

* using tobacco and alcohol one week before surgery and during the study
* dealing with mercury in their job like dentists, stonemason, mine workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Blood mercury concentration | within the 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Saatchi, DDS, MS, Study Chair — Department of Endodontics and Torabinejad Dental Research Center, School of Dentistry, Isfahan University of Medical Sciences
Locations (1):
- School of Dentistry, Isfahan University of Medical Sciences, Isfahan, Isfahan, Iran

REFERENCES:
- See also: Web Site of Isfahan University of Medical Sciences — http://mui.ac.ir/en/